CLINICAL TRIAL: NCT04326517
Title: Microbiologic Profile And Factors Associated To Intensive Care Admission And Mortality In Patients With Emphysematous Pyelonephritis: A 10-Year Experience In A Tertiary Care Center
Brief Title: Factors Associated To Intensive Care Admission And Mortality In Patients With Emphysematous Pyelonephritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Adrián Gutiérrez González, Head of Urology Department, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: UR 18-00008
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Emphysematous Pyelonephritis
Keywords: emphysematous pyelonephritis; intensive care unit; mortality; risk factors
MeSH Terms: conditions — Emphysematous Pyelonephritis | interventions — Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emphysematous pyelonephritis: This is a single-group cohort study. A sub-classification will be used in order to differentiate patients that did not require intensive care, the ones who admitted to intensive care and mortality.
  Interventions: Procedure: Nephrectomy

INTERVENTIONS:
Procedure: Nephrectomy — Different therapeutic options are described in literature for emphysematous pyelonephritis. In our center, medical treatment (no invasive procedure), ureteral stent (endourologic procedure), percutaneous drainage (minimally invasive procedure), and nephrectomy are the therapeutic options for this disease.
  Other Names: ureteral stent; percutaneous drainage; medical treatment

SUMMARY:
Emphysematous pyelonephritis is a lifethreatening necrotizing infection of the kidney characterized by accumulation of gas in the renal parenchyma and within the surrounding tissues. The aim of the study is to report the outcome of the management of this condition at the investigators institution and to determine the microbiological characteristics, antibiotic resistance patterns, and to analyze factors predicting mortality and intensive care unit admission.

DETAILED DESCRIPTION:
The investigators are planning to perform a retrospective study analyzing cases of emphysematous pyelonephritis from a single tertiary care institution in the north of Mexico in the period of 2011-2021. The diagnosis of emphysematous pyelonephritis is confirmed by computed tomography. Demographic, clinical, biochemical, therapeutic management, and outcomes will be collected. Variables will be analyzed to determine factors associated with admission to intensive care unit and mortality. Urine cultures will be analyzed and drug resistance profile will be determined using microdilution plate. Clinical and demographic characteristics will be analyzed using Chi square test for categorical variables, and T-test for numerical variables. Statistical significance is set at p<0.05. Statistical analysis will be performed with the SPSS software version 20.0.

ELIGIBILITY:
Inclusion Criteria:

* Emphysematous pyelonephritis confirmed with computed tomography
* Systemic inflammatory response
* Urinary tract infection symptoms
* Complete medical records
* Both genders included
* >18 years old

Exclusion Criteria:

* Other infectious causes
* Asymptomatic bacteriuria
* Incomplete medical records
* Endourologic procedure 3 months before recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmatory diagnosis using emphysematous pyelonephritis by computed tomography are included, as well as signs and symptoms of upper urinary tract infection and data of systemic inflammatory response. Participants are usually admitted to the emergency room and recruited for analysis during hospitalization.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with admission to Intensive care unit | 10 years
  Patients with criteria to admit to intensive care unit
Rate of mortality | 10 years
  Death cases during hospitalization

SECONDARY OUTCOMES:
Antibiotic susceptibility | 10 years
  Drug resistance profile will be determined using microdilution plate.

CONTACTS AND LOCATIONS:
Overall Officials: Adrián Gutiérrez-González, PhD, Principal Investigator — Universidad Autónoma de Nuevo León
Locations (1):
- Hospital Universitario "Dr. José Eleuterio González", Monterrey, Outside U.S./Canada, Mexico

IPD SHARING:
Plan to Share IPD: Yes
An e-mail contact of the research party will be published in order to share information of our data, excel databases and other type of information.
Supporting Information: Study Protocol, SAP
Time Frame: after recruitment period has concluded.
Access Criteria: By e-mail, any author will be available in order to support and facilitate requested information.

REFERENCES:
- [Result] Michaeli J, Mogle P, Perlberg S, Heiman S, Caine M. Emphysematous pyelonephritis. J Urol. 1984 Feb;131(2):203-8. doi: 10.1016/s0022-5347(17)50309-2. No abstract available. PMID 6366247
- [Result] Pontin AR, Barnes RD, Joffe J, Kahn D. Emphysematous pyelonephritis in diabetic patients. Br J Urol. 1995 Jan;75(1):71-4. doi: 10.1111/j.1464-410x.1995.tb07237.x. PMID 7850302
- [Result] Ubee SS, McGlynn L, Fordham M. Emphysematous pyelonephritis. BJU Int. 2011 May;107(9):1474-8. doi: 10.1111/j.1464-410X.2010.09660.x. Epub 2010 Sep 14. PMID 20840327
- [Result] Kumar A, Turney JH, Brownjohn AM, McMahon MJ. Unusual bacterial infections of the urinary tract in diabetic patients--rare but frequently lethal. Nephrol Dial Transplant. 2001 May;16(5):1062-5. doi: 10.1093/ndt/16.5.1062. No abstract available. PMID 11328918
- [Result] Huang JJ, Tseng CC. Emphysematous pyelonephritis: clinicoradiological classification, management, prognosis, and pathogenesis. Arch Intern Med. 2000 Mar 27;160(6):797-805. doi: 10.1001/archinte.160.6.797. PMID 10737279
- [Result] Falagas ME, Alexiou VG, Giannopoulou KP, Siempos II. Risk factors for mortality in patients with emphysematous pyelonephritis: a meta-analysis. J Urol. 2007 Sep;178(3 Pt 1):880-5; quiz 1129. doi: 10.1016/j.juro.2007.05.017. Epub 2007 Jul 16. PMID 17631348
- [Result] Huang JJ, Chen KW, Ruaan MK. Mixed acid fermentation of glucose as a mechanism of emphysematous urinary tract infection. J Urol. 1991 Jul;146(1):148-51. doi: 10.1016/s0022-5347(17)37736-4. PMID 2056576
- [Result] Somani BK, Nabi G, Thorpe P, Hussey J, Cook J, N'Dow J; ABACUS Research Group. Is percutaneous drainage the new gold standard in the management of emphysematous pyelonephritis? Evidence from a systematic review. J Urol. 2008 May;179(5):1844-9. doi: 10.1016/j.juro.2008.01.019. Epub 2008 Mar 19. PMID 18353396